CLINICAL TRIAL: NCT04743778
Title: Online Diabetes Education Project: Virtual Diabetes Self-Management Education and Support Intervention
Brief Title: Online Diabetes Education Project (ODEP)
Acronym: ODEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jaclynn Hawkins, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODEP HUM00190508; P30DK092926 (NIH)
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Initially, we intended to have a control group and an intervention group. However, due to low recruitment numbers and COVID-19 pandemic barriers, we decided to offer all participants virtual DSME/S.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Diabetes Self-Management Education and Support (Experimental): Participants will receive one hour of DSME/S delivered by a Certified Diabetes Care and Education Specialist (CDCES) per week for 10 weeks delivered via the Zoom for Health at U-M service may be used for Protected Health Information (PHI, regulated by HIPAA). To ensure treatment fidelity, three DSME/S sessions will be selected at random and recorded and rated for fidelity to the above content by our research team.
  Interventions: Behavioral: Virtual Diabetes Self-Management Education and Support

INTERVENTIONS:
Behavioral: Virtual Diabetes Self-Management Education and Support — Diabetes self-management education and support delivered through Zoom for health.

SUMMARY:
This pilot randomized control trial will be testing an empowerment-based virtual group diabetes self-management education and support (DSME/S) for African American/Black adults with type 2 diabetes living in Detroit. Participants will be randomized to either a control group or the virtual DSME/S group.

DETAILED DESCRIPTION:
This pilot randomized control trial will be testing an empowerment-based virtual group diabetes self-management education and support (DSME/S) for African American/Black adults with type 2 diabetes living in Detroit. Participants interested in participating in this study will first be consented then they will complete a baseline health assessment including a questionnaire and physiologic testing. Using a 50/50 randomization scheme, participants will be randomized to either a control group or the virtual DSME/S group and be told of their placement. Participants randomized to the control group will receive community resources, diabetes specific newsletters, and pedometers. Participants randomized to the virtual DSME/S group will receive 10-weekly 1-hour virtual DSME/S sessions with a certified diabetes care and education specialists through Zoom for Health at the University of Michigan, a HIPPA compliant platform. After the intervention is complete and then again 3 months later, participants in both groups will be invited to complete an additional health assessment.

However, due to low recruitment we removed the control arm and offered all participants virtual DSME/S.

ELIGIBILITY:
Inclusion Criteria:

* Agee 18 or older, Black, a diagnosis of T2D for one year duration or longer, ambulatory status.

Exclusion Criteria:

* Non-ambulatory, serious health conditions (morbid obesity and severe symptomatic heart disease, visual impairment, renal failure, and peripheral neuropathy), psychiatric illness (severity requiring hospitalization) or cognitive deficit (illness determined using the Montreal Cognitive Assessment tool) and serious diabetes complications (e.g. blindness) that would impede meaningful participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclynn Hawkins, MSW, PhD, Principal Investigator — University of Michigan, School of Social Work
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Diabetes Self-Management Education and Support
Started | 12
Completed | 8
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Control of A1c (Mean Change in A1C)
Description: Measured using the DCA 2000 point-of-care testing instrument. The American Diabetes Association recommends people living with diabetes to have an A1C below 7.0%.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
percent | -0.02 (1.64)

2. Primary Outcome: Depression
Description: Measured using the Patient Health Questionnaire (PHQ-9). A PHQ-9 score of 0-4 means none-minimal depression severity, a score of 5-9 means mild depression severity, a score of 10-14 means moderate depression severity, a score of 15-19 means moderately severe depression, and 20-27 means severe depression.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
units on a scale | -0.79 (4.14)

3. Primary Outcome: Regimen Adherence
Description: Measured using the Perceived Diabetes Self-Management Scale (PDSMS), a self-report questionnaire used to measure a broad range of management behaviors, such as insulin management, dietary management, blood glucose monitoring, symptom response, and parent assistance/supervision. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes. For this study, we reported mean change in PDSMS score.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
units on a scale | 1.12 (4.01)

4. Secondary Outcome: Body Mass Index (BMI)
Description: Calculated using height and weight. Height will be measured using a stadiometer. Weight will be measured on a high quality, calibrated digital scale. Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9 Obesity = BMI of 30 or greater
  For this study, we reported the mean change in BMI.
Time Frame: baseline 3 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
kg/m^2 | -0.54 (10.34)

5. Secondary Outcome: Blood Pressure
Description: Measured using the auscultatory method. The American Diabetes Association recommends people living with type 2 diabetes to have a blood pressure target of 130/80 mmHg.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
mmHg
  Systolic | 7.75 (14.75)
  Diastolic | 5.33 (10.76)

6. Secondary Outcome: Diabetes Social Support
Description: Measured using the Chronic Illness Resources Survey. This survey has a minimum score of 22 and a maximum score of 110. The higher the value, the more support and resources someone has for managing their illness. We measured the mean change in score.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
units on a scale | 0.48 (1.23)

7. Secondary Outcome: Diabetes-Related Distress
Description: Measured using the Diabetes Distress Scale. The score is calculated by averaging 17 items on the questionnaire. Scores range from 1 to 6, with 1 being the least distressed and 6 being the most distressed. We consider a mean item score of 3 or higher (moderate distress) as a level of distress worthy of clinical attention. We reported the mean change in diabetes distress below.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Virtual Diabetes Self-Management Education and Support: Participants randomized into the virtual empowerment-based DSME/S group will receive one hour of DSME/S delivered by a Certified Diabetes Care and Education Specialist (CDCES) per week for 10 weeks delivered via the Zoom for Health at U-M service may be used for Protected Health Information (PHI, regulated by HIPAA). To ensure treatment fidelity, three DSME/S sessions will be selected at random and recorded and rated for fidelity to the above content by our research team.
  Virtual Diabetes Self-Management Education and Support: Diabetes self-management education and support delivered through Zoom for health.
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
units on a scale | -5.72 (14.46)

8. Secondary Outcome: Diabetes Quality of Life
Description: Measured using the Diabetes Quality of Life Questionnaire. The 46-item DQoL scale consists of four domains and is measured using a 5-point Likert scale, where scores are averaged across all domains and summed. Scores range from 0 to 100. The higher the score, the higher the quality of life. We reported the mean change below.
Time Frame: baseline and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Diabetes Self-Management Education and Support
Number analyzed (Participants) | 12
units on a scale | 0.14 (0.65)

ADVERSE EVENTS:
Time Frame: 3 months (duration of study)
Arm/Group | Virtual Diabetes Self-Management Education and Support
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT04743778/Prot_SAP_000.pdf